CLINICAL TRIAL: NCT02900482
Title: Research for Genetic Factors Involved in Congenital Dislocation of Hip: Genome-wide Association Study in Grand West France
Acronym: GENETHIP
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: RB 11.042 GENETHIP
Record Dates: First submitted 2016-08-26; First posted 2016-09-14 (Estimated); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Congenital Hip Dislocation
MeSH Terms: conditions — Hip Dislocation, Congenital

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- case group: Patients with a history of congenital hip dislocation
  Interventions: Other: Sampling saliva
- control group: Patients with no history of congenital hip dislocation
  Interventions: Other: Sampling saliva
- parents of case group: Parents of patients with a history of congenital hip dislocation
  Interventions: Other: Sampling saliva

INTERVENTIONS:
Other: Sampling saliva

SUMMARY:
The main objective is to identify the genes involved in congenital dislocation of the hip.

The secondary objectives are to measure the association between mechanical risk factors and congenital dislocation of hip and study the interactions between these factors and genetic factors.

DETAILED DESCRIPTION:
Congenital hip dislocation (CHD) is one of the most frequent skeleton abnormalities in the Caucasian population (incidence: 2-10 / 1000). This disease results from an abnormality of the reports of the femoral head with the acetabulum, generated by a morphological defect of the cavity and / or joint hypermobility.

This condition is now defined as a multifactorial disease involving in the one hand, mechanical factors related to the conditions of pregnancy and childbirth, and secondly, genetic factors suggested by ethnic predisposition and familial aggregation observed. Despite the neonatal screening, CHD remains a public health problem because of its high frequency, because of the functional handicap which it leads in case of late diagnosis and of its natural evolution to coxarthrosis.

CHD was the object of a significant number of publications on the difficult aspects of its screening and treatment but, at the moment, few data are available on the genetic factors involved.

The genetic studies led on the CHD based on studies of case-control associations, focused on candidate genes, and genetic linkage analysis, two strategies classically used in genetic epidemiology.

To date, these strategies did not allow to elucidate the genetic determinism of the pathology.

The considerable progress made in recent years both in the field of knowledge of the human genome and its variability, in the development of methodological and technological tools allow to better understand the genetic determinism of complex diseases such as CHD.

The development of the techniques of broadband sequencing, new generation said sequencing (NGS for Next Generation Sequencing) makes indeed accessible the sequencing of the whole genome or of the set of its coding regions (exome) and now allows identify rare variants, that is to say variants having a minor allele frequency of less than 1%. These variants were previously not recognizable by the strategies traditionally used in genetic epidemiology, which are based on the study of common variants (minor allele frequency of ≥ 5%) listed in the public databases of the human genome .

The NGS sequencing technique makes it possible to address the problem of the study of complex diseases in a new light and it appears necessary to apply this strategy to the CHD to search for genetic factors involved in the pathology.

The genetic analysis strategy initially envisaged consisted of a genome wide association study (GWAS), which aims to genotype millions of frequent genetic markers scattered along the genome and to test their association with the disease.

The technological advances made in the field of molecular genetics since the implementation of the GENETHIP protocol have made it possible to envisage new strategies to identify the genetic factors involved in a complex disease such as CHD. These strategies include high-throughput sequencing - Next Generation Sequencing (NGS) - which now makes sequencing of all coding regions of the genome (exome) possible. Beyond the frequent variants, this technique also makes it possible to identify rare variants (frequency of the minor allele <1%), not analyzed by the strategy initially envisaged in this project.

It was therefore decided to adopt this new strategy in the GENETHIP study. The sample size could be reduced as the average frequency of the minor allele is lower with this type of study.

The new genetic strategy adopted nevertheless requires the inclusion of selected phenotypes, which leads to recruiting exclusively patients with a family history of congenital hip disorders and excluding those who have had a presentation by the seat (main mechanical risk factor of the CHD). This is intended to better target the genetic character of the pathology.

ELIGIBILITY:
Inclusion Criteria:

* Old patient at least of 3 weeks and under age 16 presenting a congenital pathology of hip defined by the following consensual criteria:

  1. Ultrasound criteria: osseous Cover of the femoral head 50 % or Bottom cotyloïdien = 6 mm or Type III and IV of the classification of Graf
  2. Radiographic criteria: acetabular angle = 30 ° or Absence of projection of the femoral pit in the infero-internal quadrant of the construction of Ombredanne or acetabular angle upper of more than 5 ° with regard to the healthy side (so reached unilateral)
* Patient presenting family history of congenital hip dislocation
* Patient of Caucasian origin
* Signature of the consent

Exclusion Criteria:

* Patient presenting anomalies of the collagen and/or the elastic tissue ( imperfect osteogenesis, syndromes of Ehlers-Danlos, Larsen and Marfan)
* Patient presenting karyotype abnormalities
* Refusal to participate

Ages: 3 Weeks to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Case group
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2012-11-23 (Actual); Primary Completion 2022-11-03 (Actual); Study Completion 2022-11-03 (Actual)

PRIMARY OUTCOMES:
Research for one or several genes involved in the congenital dislocation of hip by comparing the DNA from blood or saliva of patients and controls. | inclusion
  The primary endpoint of the study is to sequence exome of patients affected by congenital dislocation of hip and of controls to identify one or several genes involved in the congenital dislocation of hip and compare the distribution of variants identified by exome sequencing between patients and controls.

CONTACTS AND LOCATIONS:
Locations (1):
- Bertrand Fenoll, Brest, France

IPD SHARING:
Plan to Share IPD: No